CLINICAL TRIAL: NCT01143194
Title: A Randomized, Placebo-Controlled, Double-Blind, Crossover Study to Evaluate the Effects of Three Doses of the Dietary Supplement oréVida™ on Alertness, Attention and Concentration in Healthy Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Kathleen Kelley, MD, Provident Clinical Research and Consulting,Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2009-11-06-OREG
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Attention; Memory; Alertness
Keywords: Attention; Vigilance; Concentration; Memory; Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- oréVida™ 60mg/day (Experimental)
  Interventions: Dietary Supplement: oréVida™
- oréVida™ 120mg/day (1) (Experimental)
  Interventions: Dietary Supplement: oréVida™
- oréVida™ 120mg/day (2) (Experimental)
  Interventions: Dietary Supplement: oréVida™
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: oréVida™ — 1 capsule 30 mg oréVida™ twice a day (one in the morning, one in the afternoon, so in total 60 mg/day)
  Arms: oréVida™ 60mg/day
Dietary Supplement: oréVida™ — 1 capsule 60 mg oréVida™ twice a day (one in the morning, one in the afternoon, so in total 120mg/day)
  Arms: oréVida™ 120mg/day (1)
Dietary Supplement: oréVida™ — 1 capsule 120 mg oréVida™ in the morning, one placebo capsule in the afternoon (si in total 120 mg/day)
  Arms: oréVida™ 120mg/day (2)
Dietary Supplement: Placebo — 1 capsule of placebo twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of the dietary supplement oréVida™ (active ingredient on the basis of a culinary herb)administered twice daily in an acute study on an improvement in vigilance, attention, concentration, memory and mood in 45 healthy men and pre-menopausal women, aged 35-50 years, inclusive.

oréVida™ is considered a dietary supplement, and therefore it is not an approved drug by the Food and Drug Administration (FDA). It is regulated like a food. The U.S. Food and Drug Administration does not strictly regulate herbs and dietary supplements. We do not claim that this supplement is meant to treat any ailment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or pre-menopausal female, 35-50 years, inclusive. Post-menopausal is defined as a history of spontaneous amenorrhea for a period of 12 consecutive months or six weeks post-surgical bilateral oophorectomy, with or without hysterectomy.
* Subject is willing to maintain his or her habitual diet and usual physical activity patterns throughout the study.
* Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
* Subject has a body mass index (BMI) of ≥20.00 and <30.00 kg/m2
* Subject is willing to refrain from consuming alcohol 24 h prior to test days.
* Subject is willing to refrain from consuming caffeine and caffeine-containing products 12 h prior to test days.
* Subject is willing to refrain from vigorous physical activity 12 h prior to test days.
* Subject is a non-smoker.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Subject has a positive drug screening of amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, methamphetamines, methadone, 3,4-methylenedioxymethamphetamine, opiates or tricyclic antidepressants at screening.
* Subject has abnormal laboratory test results of clinical significance, including, but not limited to: creatinine ≥1.5 mg/dL, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥1.5X the upper limit of normal at screening.
* Subject has donated more than 300 mL of blood during the three months prior to screening.
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the average blood pressure measured at screening. One re-test will be allowed on a separate day prior to visit 2, day 0 for subjects whose blood pressure exceeds either of these cut points at visit 1.
* Subject has a history or presence of clinically important cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorders that, in the judgment of the Investigator, would interfere with the subject's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the subject at undue risk.
* Subject has a history, in the judgment of the Investigator, of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Use of any sleep aid medication within four days prior to each test day.
* Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
* Subject is pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
* Excessive habitual caffeine consumption (>300 mg caffeine/d or ≥3 cups of caffeinated coffee/d), following screening and throughout the study period.
* Use of any psychotropic medication within four weeks of screening and throughout the study.
* Use of antibiotics or signs of active systemic infection. Treatment visits will be rescheduled to allow the subject to wash off of the antibiotic for at least five days prior to any test visit.
* Subject has had exposure to any non-registered drug product within 30 days prior to the screening visit.
* Use of dietary supplements containing any of the following: ginkgo biloba, St. John's wort, ginseng, gotu kola (Indian pennywort); daily doses of vitamin E (≥30 mg/d) or folic acid (≥400 ug/d); thiamine, riboflavin, and/or pyridoxine (≥2 mg/d); and eicosapentaenoic acid (EPA), docosahexaenoic acid or a combination of EPA + DHA (≥500 mg/d) within 2 weeks of screening visit.
* Recent history of (within 12 months of screening visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Subject has a known allergy or sensitivity to study product or any ingredients of the study product or meals provided.
* The subject is unable to perform the tests on the CDR System during training to the established acceptable levels for participation in this type of study.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Vigilance, Attention, and Concentration Tasks | 4 times one day (at each test day, tasks 13 times repeated)
  Cognitive Drug Research (CDR) Test Battery Attention:
  * Simple Reaction Time (Speed (msec))
  * Digit Vigilance (Speed (msec)/ Targets detected (%))
  * Choice Reaction Time(Speed (msec))

SECONDARY OUTCOMES:
Working Memory & Executive Function Tasks | 4 times one day (at each test day, tasks 7 times repeated)
  CDR Test Battery Memory:
  * Numeric Working Memory (Sensitivity (SI); Speed (msec))
  * Spatial Working Memory (Sensitivity (SI); Speed (msec))
Episodic Secondary Memory Tasks | 4 times one day (at each test day, tasks 7 times repeated)
  CDR Test Battery Memory:
  * Immediate Word Recall (Words correctly recalled (%))
  * Delayed Word Recall (Words correctly recalled (%)
  * Word Recognition (Sensitivity (SI); Speed (msec))
  * Picture Recognition (Sensitivity (SI); Speed (msec))
Additional Measurements / Questionnaires | 4 times one day (at each test day, VAS 13 times repeated / POMS 3 times repeated)
  * Bond-Lader Visual Analog Scale (VAS) of Mood and Alertness
  * Profile of Mood States (POMS) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kelley, MD, Principal Investigator — Provident Clinical Research
Locations (1):
- Provident Clinical Research, Addison, Illinois, United States